CLINICAL TRIAL: NCT05325476
Title: Testing of the JomPrEP App for HIV Prevention Among Malaysian MSM
Acronym: JomPrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: University of Malaya (Other); National Institutes of Health (NIH) (NIH); Yale University (Other)
Responsible Party: Principal Investigator, Roman Shrestha, Assistant Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R33TW011665 (NIH)
Record Dates: First submitted 2022-03-24; First posted 2022-04-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: HIV Prevention Program
Keywords: PrEP; mHealth; Smartphone app; mobile app; men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JomPrEP App Group (Experimental): Participants in the TAU group will receive the JomPrEP app with major intervention features inactivated; information and resources for HIV testing, PrEP, and available mental health and addiction services will be available along with access to risk assessment tools. The Research Assistant will assist in downloading the app and provide a tutorial in using the assessment tool of the app.
  Interventions: Other: JomPrEP App
- Treatment as usual (Active Comparator): Participants in the JomPrEP group will be provided with full app access. The Research Assistant will use an onboarding checklist to orient participants to download the app and its use. Participants will be encouraged to explore and use all components of the app. Participants will be able to personalize the frequency, timing, and content for daily adherence support and weekly behavioral feedback messages and receive reminders for regular PrEP care. Participants can also contact the Research Assistant using the chat function for support and assistance with linkage to services.
  Interventions: Other: Inactivated JomPrEP app

INTERVENTIONS:
Other: JomPrEP App — The JomPreP app will be ideally designed to optimize HIV prevention cascade by providing a virtual platform to access to HIV prevention (e.g., HIV testing and PrEP) and other support services (e.g., mental health). The JomPrEP app will be available on the Apple Store and the Google Play Store for the users to download. However, access to the app will be restricted to the research participant using a unique registration code.
  Arms: JomPrEP App Group
Other: Inactivated JomPrEP app — Participants will have access to the JomPrEP app with major intervention features inactivated. Information and resources for HIV testing, PrEP, and available mental health and addiction services will be available along with access to risk assessment tools. The RA will assist in downloading the app and provide a tutorial in using the assessment tool of the app.
  Arms: Treatment as usual

SUMMARY:
This project will involve conducting a Type I Hybrid Implementation Science trial to assess the efficacy of the JomPrEP app while measuring contextual implementation factors to guide its future adoption and scale-up.

DETAILED DESCRIPTION:
mHealth is a promising and cost-effective strategy to reach stigmatized and hard-to-reach populations, like MSM, and link them to care. Leveraging mHealth reduces individuals' discomfort and distrust of disclosing risk behaviors to providers, providers' low cultural competency for working with individuals of diverse sexual identities, and bypasses barriers to health care for marginalized populations, - all features crucial for HIV prevention in MSM in Malaysia. It can further guide prevention delivery and health decision-making in a confidential, less stigmatizing, and convenient manner.

Results from our studies show Malaysian MSM often do not get HIV tested, initiate PrEP, or have their mental health needs addressed. Mixed methods suggest MSM want these services but prefer a streamlined system to access them that reduces interaction with clinicians where disclosure and perceived judgment occurs. mHealth may overcome these barriers by doing the screening confidentially and result in an "eligibility" output that automates HIV prevention service delivery (e.g., HIV testing, pre-exposure prophylaxis; PrEP). Overall smartphone growth in Malaysia (63% in 2015 to 89% in 2017) and our parallel work with MSM indicates that nearly all (>97%) MSM own a smartphone; Internet penetration is 89.4%, mostly through smartphones. Findings from our qualitative interviews with MSM further indicate stated preferences for interfacing with 'apps' rather than health professionals to access HIV testing, PrEP, counseling, and sexual health services as well as stakeholders indicating strong interest in using app-based platforms to deliver integrated care (e.g., HIV, mental health) align with developing culturally tailored mHealth strategies and to engage MSM in virtual communication with providers about their unmet needs for HIV testing, PrEP, and mental and sexual needs - all embedded within one app. The cross-cutting prevention strategies like the use of mHealth, particularly smartphone apps, thus hold great promise for HIV prevention in Malaysian MSM, especially when linked to HIV testing, PrEP, and co-morbid P/SUD screening and feedback, which will likely facilitate adherence and reduce HIV risk.

Although mHealth has been widely applied and efficacious in promoting health outcomes in multiple patient populations and contexts, app-based platforms to improve the HIV prevention cascade are just emerging. Few apps specifically to increase uptake and adherence to PrEP are evolving and limited to high-income countries. Further, these apps do not address mental health issues that are common in those who need HIV prevention most.

Given the evolving HIV epidemic among men who have sex with men (MSM) in Malaysia and their challenges with accessing prevention services, we previously proposed to adapt, expand, and refine an existing app (namely the HealthMindr app) to deliver an integrated HIV prevention intervention that will promote HIV testing and linkage to pre-exposure prophylaxis (PrEP) and that incorporates screening and support for psychiatric and substance use disorder (P/SUD) for Malaysian MSM. We have previously developed a new app (called JomPrEP) designed to improve access to HIV prevention services (i.e., HIV testing and PrEP) among Malaysian MSM. We now plan to conduct a Type 1 Hybrid Implementation Science Trial to (1) evaluate the efficacy of the JomPrEP app vs. treatment as usual (TAU) in Malaysian MSM (using a randomized controlled trial) and (2) assess contextual implementation factors (using focus groups).

ELIGIBILITY:
Inclusion Criteria:

* HIV negative or status unknown
* Cis-gender men who have sex with men
* Age more than or equal to 18 years
* Own a smartphone (Android or IOS)

Exclusion Criteria:

* Unable to read or understand English or Bahasa Malaysia
* Unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender men
Enrollment: 268 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Changes in HIV testing | 3, 6, and 9 months post-randomization
  HIV testing dates will be assessed at each follow-up time point (3, 6, and 9 months) using self-report.
Changes in PrEP uptake | 3, 6, and 9 months post-randomization
  PrEP uptake (current use of PrEP; yes/no) will be assessed at each follow-up time point (3, 6, and 9 months) using self-reported visual analogue scale. The higher the score on the scale the higher the PrEP uptake. Score (0-100).

SECONDARY OUTCOMES:
Changes in PrEP adherence | 3, 6, and 9 months post-randomization
  PrEP Adherence will be assessed using Dried Blood Spots at 3-, 6-, and 9-month follow-ups, which will quantify tenofovir-diphosphate (TFV-DP) and emtricitabine-triphosphate (FTC-TP) in RBC.TFV-DP ≥700 fmol/punch will be defined as optimal adherence.

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - CERiA, Kuala Lumpur
  - University of Malaya, Kuala Lumpur

REFERENCES:
- [Background] Cooper V, Clatworthy J, Whetham J, Consortium E. mHealth Interventions To Support Self-Management In HIV: A Systematic Review. Open AIDS J. 2017 Nov 21;11:119-132. doi: 10.2174/1874613601711010119. eCollection 2017. PMID 29290888
- [Background] Henny KD, Wilkes AL, McDonald CM, Denson DJ, Neumann MS. A Rapid Review of eHealth Interventions Addressing the Continuum of HIV Care (2007-2017). AIDS Behav. 2018 Jan;22(1):43-63. doi: 10.1007/s10461-017-1923-2. PMID 28983684
- [Background] Conserve DF, Jennings L, Aguiar C, Shin G, Handler L, Maman S. Systematic review of mobile health behavioural interventions to improve uptake of HIV testing for vulnerable and key populations. J Telemed Telecare. 2017 Feb;23(2):347-359. doi: 10.1177/1357633X16639186. Epub 2016 Jul 9. PMID 27056905
- [Background] Marcolino MS, Oliveira JAQ, D'Agostino M, Ribeiro AL, Alkmim MBM, Novillo-Ortiz D. The Impact of mHealth Interventions: Systematic Review of Systematic Reviews. JMIR Mhealth Uhealth. 2018 Jan 17;6(1):e23. doi: 10.2196/mhealth.8873. PMID 29343463
- [Background] WHO. mHealth: New horizons for health through mobile technologies: second global survey on eHealth. Geneva, Switzerland2011.
- [Background] Free C, Phillips G, Watson L, Galli L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technologies to improve health care service delivery processes: a systematic review and meta-analysis. PLoS Med. 2013;10(1):e1001363. doi: 10.1371/journal.pmed.1001363. Epub 2013 Jan 15. PMID 23458994
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Background] Milward J, Lynskey M, Strang J. Solving the problem of non-attendance in substance abuse services. Drug Alcohol Rev. 2014 Nov;33(6):625-36. doi: 10.1111/dar.12194. Epub 2014 Sep 6. PMID 25196817
- [Background] Mbuagbaw L, Mursleen S, Lytvyn L, Smieja M, Dolovich L, Thabane L. Mobile phone text messaging interventions for HIV and other chronic diseases: an overview of systematic reviews and framework for evidence transfer. BMC Health Serv Res. 2015 Jan 22;15:33. doi: 10.1186/s12913-014-0654-6. PMID 25609559
- [Background] Chawarski MC, Vicknasingam B, Mazlan M, Schottenfeld RS. Lifetime ATS use and increased HIV risk among not-in-treatment opiate injectors in Malaysia. Drug Alcohol Depend. 2012 Jul 1;124(1-2):177-80. doi: 10.1016/j.drugalcdep.2011.12.024. Epub 2012 Jan 21. PMID 22266088
- [Background] Fendrich M, Avci O, Johnson TP, Mackesy-Amiti ME. Depression, substance use and HIV risk in a probability sample of men who have sex with men. Addict Behav. 2013 Mar;38(3):1715-8. doi: 10.1016/j.addbeh.2012.09.005. Epub 2012 Sep 24. PMID 23254224
- [Background] Daskalopoulou M, Rodger A, Phillips AN, Sherr L, Speakman A, Collins S, Elford J, Johnson MA, Gilson R, Fisher M, Wilkins E, Anderson J, McDonnell J, Edwards S, Perry N, O'Connell R, Lascar M, Jones M, Johnson AM, Hart G, Miners A, Geretti AM, Burman WJ, Lampe FC. Recreational drug use, polydrug use, and sexual behaviour in HIV-diagnosed men who have sex with men in the UK: results from the cross-sectional ASTRA study. Lancet HIV. 2014 Oct;1(1):e22-31. doi: 10.1016/S2352-3018(14)70001-3. Epub 2014 Sep 7. PMID 26423813
- [Background] Hirshfield S, Remien RH, Humberstone M, Walavalkar I, Chiasson MA. Substance use and high-risk sex among men who have sex with men: a national online study in the USA. AIDS Care. 2004 Nov;16(8):1036-47. doi: 10.1080/09540120412331292525. PMID 15511735
- [Background] Van Tieu H, Koblin BA. HIV, alcohol, and noninjection drug use. Curr Opin HIV AIDS. 2009 Jul;4(4):314-8. doi: 10.1097/COH.0b013e32832aa902. PMID 19532070
- [Background] Halkitis PN, Parsons JT. Recreational Drug Use and HIV-Risk Sexual Behavior Among Men Frequenting Gay Social Venues. Journal of Gay & Lesbian Social Services. 2002;14(4):19-38.
- [Background] Sandfort TGM, Knox JR, Alcala C, El-Bassel N, Kuo I, Smith LR. Substance Use and HIV Risk Among Men Who Have Sex With Men in Africa: A Systematic Review. J Acquir Immune Defic Syndr. 2017 Oct 1;76(2):e34-e46. doi: 10.1097/QAI.0000000000001462. PMID 28903126
- [Background] Shrestha R, Lim SH, Altice FL, Copenhaver M, Wickersham JA, Saifi R, Ab Halim MA, Naning H, Kamarulzaman A. Use of Smartphone to Seek Sexual Health Information Online Among Malaysian Men Who Have Sex with Men (MSM): Implications for mHealth Intervention to Increase HIV Testing and Reduce HIV Risks. J Community Health. 2020 Feb;45(1):10-19. doi: 10.1007/s10900-019-00713-x. PMID 31375976
- [Background] Shrestha R, Lim SH, Altice FL, Kamarulzaman A, Wickersham J. Perception and acceptability of mHealth-based intervention for HIV prevention among men who have sex with men (MSM) in Malaysia. In preparation. 2019.
- [Background] Malaysian Communications and Multimedia Commission. Internet users survey: 2017. 2017; https://mcmc.gov.my/skmmgovmy/media/General/pdf/HPUS2017.pdf. Accessed May 1, 2019.
- [Background] Sharpe JD, Kamara MT. A systematic evaluation of mobile apps to improve the uptake of and adherence to HIV pre-exposure prophylaxis. Sex Health. 2018 Nov;15(6):587-594. doi: 10.1071/SH18120. PMID 30347177
- [Background] Biello KB, Marrow E, Mimiaga MJ, Sullivan P, Hightow-Weidman L, Mayer KH. A Mobile-Based App (MyChoices) to Increase Uptake of HIV Testing and Pre-Exposure Prophylaxis by Young Men Who Have Sex With Men: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 7;8(1):e10694. doi: 10.2196/10694. PMID 30617042
- [Background] Liu A, Coleman K, Bojan K, Serrano PA, Oyedele T, Garcia A, Enriquez-Bruce E, Emmanuel P, Jones J, Sullivan P, Hightow-Weidman L, Buchbinder S, Scott H. Developing a Mobile App (LYNX) to Support Linkage to HIV/Sexually Transmitted Infection Testing and Pre-Exposure Prophylaxis for Young Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Jan 25;8(1):e10659. doi: 10.2196/10659. PMID 30681964
- [Background] LeGrand S, Knudtson K, Benkeser D, Muessig K, Mcgee A, Sullivan PS, Hightow-Weidman L. Testing the Efficacy of a Social Networking Gamification App to Improve Pre-Exposure Prophylaxis Adherence (P3: Prepared, Protected, emPowered): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Dec 18;7(12):e10448. doi: 10.2196/10448. PMID 30563818
- [Background] Sullivan PS, Driggers R, Stekler JD, Siegler A, Goldenberg T, McDougal SJ, Caucutt J, Jones J, Stephenson R. Usability and Acceptability of a Mobile Comprehensive HIV Prevention App for Men Who Have Sex With Men: A Pilot Study. JMIR Mhealth Uhealth. 2017 Mar 9;5(3):e26. doi: 10.2196/mhealth.7199. PMID 28279949
- [Derived] Shrestha R, Wickersham JA, Khati A, Azwa I, Ni Z, Kamarulzaman A, Sullivan PS, Jadkarim L, Eger WH, Gautam K, Altice FL. Clinic-Integrated Mobile Health Intervention ("JomPrEP" App) to Improve Uptake of HIV Testing and Pre-exposure Prophylaxis Among Men Who Have Sex With Men in Malaysia: Protocol for an Intervention Development and Multiphase Trial. JMIR Res Protoc. 2022 Dec 21;11(12):e43318. doi: 10.2196/43318. PMID 36542425